CLINICAL TRIAL: NCT03663426
Title: Randomized Controlled Trial Study in Hip Arthroplasty by Direct Anterior Approach Using Opioid Free Anesthesia (OFA) Versus Standard Opioid Anesthesia.
Brief Title: Impact of Opioid Free Anesthesia on Outcome After Hip Arthroplasty by Direct Anterior Approach.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, head of dep anesthesia & intensive care, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT impact OFA on THP
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Hip Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group opioid anesthesia (Active Comparator): standard anesthesia using opioids
  Interventions: Procedure: control
- study group opioid free anesthesia (Experimental): opioid free anesthesia and high dose glucocorticoids
  Interventions: Procedure: study group

INTERVENTIONS:
Procedure: study group — 1. High dose corticoids pre-operative and 24h postoperative
  2. Opioid free general anesthesia
  3. Avoid opioids post-operative by continue clonidine, ketamine and lidocaine, only exceptional opioids after NSAID and paracetamol.
  Arms: study group opioid free anesthesia
Procedure: control — 1. No corticoids pre-operative.
  2. Opioid anesthesia
  3. Opioids post-operative after NSAID and paracetamol.
  Arms: control group opioid anesthesia

SUMMARY:
all patients with a first anterior arthroplasty, give their informed consent to be randomized to control or study protocol.

control means no high steroid dose, opioids for anesthesia; paracetamol, NSAIDs and opioids as analgesia.

study protocol means methylprednisolone 125 mg and opioid free anesthesia followed by paracetamol, NSAIDs and if needed opioids as escape.

DETAILED DESCRIPTION:
study group means for Anesthesia:

1. High dose corticoids pre-operative: 125 mg Methylprednisolone. (Medrol) pre incision and 24h postoperative
2. OFA using a multimodal approach including alpha2agonists, lidocaine and low dose ketamine (max 1mg/kg).
3. Avoid opioids post-operative by using multimodal non-opioid analgesics after OFA. Avoid epidural to allow rapid mobilization.

all patients get Tranexamic acid 1 g (2 amp Exacyl 500mg) before and 1 g after surgery. It act as antifibrinolytic to reduce postoperative bleeding. (reversibly binding to lysine receptor sites on plasminogen) Try to give Continuous deep neuromuscular block (NMB) with a post titanic count (PTC) < 3 by continuous infusion and monitoring of NMB.

Intravenous Fluid restrictions to 1 ml/kg/h as long as pulse pressure (or plethysmograph) variation < 20% to reduce wound edema.

The pericapsular injections of local anesthetic, provided the patient had no contraindications such as poor renal function or allergies. 100 ml Ropivacaine 0,2% (max dose 3 mg/kg) + additives (Adrenaline 2,5 cc) (Ropivacaine: max 3 mg/kg)

ELIGIBILITY:
Inclusion Criteria:

* arthroplasty by anterior approach

Exclusion Criteria:

* allergy or impossible to use any of the drugs included
* revision procedure
* major cardiovascular, pulmonary or renal insufficiency requiring planned post operative intensive care admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
QoR15 | measured at 24 hours after surgery.
  quality of recovery (QoR15) measured by 15 questions evaluating condition of recovery) scale 0 to 15 with 0 being very bad while 15 being maximum recovery possible or equal to pre operative state.
opioids postoperative | measured at 24 hours after surgery.
  opioid use postoperative at 24 hours
CRP | measured at 24 hours after surgery.
  Chronic reactive protein (CRP) change 24 h post-operative

SECONDARY OUTCOMES:
surgical condition | after surgery
  surgeon scores the surgical conditions on an adapted five-point Leyden scale
muscle damage | after surgery
  surgeon scores the muscle damage on an adapted five-point Leyden scale
length of hospital stay | until hospital discharge, maximum 7 days after surgery.
  number days patient stay in the hospital before discharge
complications | 2 weeks postoperative
  complications up to two weeks postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Marco Lanckneus, MD, Study Director — AZSint Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No